CLINICAL TRIAL: NCT00642616
Title: A Phase 3, Open-label, Randomized Clinical Trial to Evaluate the Safety of Technosphere® Insulin Inhalation Powder in Type 1 or Type 2 Diabetic Subjects With Obstructive Pulmonary Disease (Asthma or Chronic Obstructive Pulmonary Disease) Over a 12 Months Treatment Period With a 2 Month Follow-up
Brief Title: Evaluate Safety of Technosphere® Insulin (TI) in Diabetic Subjects With Moderate Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated upon recommendation of the Data Safety Monitoring Board (DSMB)
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-134
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Moderate Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Asthma | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Technosphere® Insulin (Asthma) (Experimental): Technosphere® Insulin Inhalation Powder administered prandially in diabetic participants with Asthma
  Interventions: Drug: Technosphere® Insulin
- Usual Care (Asthma) (Active Comparator): Usual anti diabetic care in Diabetic participants with Asthma
  Interventions: Drug: Usual Care
- Technosphere® Insulin (COPD) (Experimental): Technosphere® Insulin Inhalation Powder administered prandially in diabetic participants with Chronic Obstructive Pulmonary disease (COPD)
  Interventions: Drug: Technosphere® Insulin
- Usual Care (COPD) (Active Comparator): Usual anti diabetic care in Diabetic participants with Chronic Obstructive Pulmonary disease (COPD)
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Technosphere® Insulin — Technosphere® Insulin delivered with Gen 2 inhaler with doses individualized for each participant in combination with an antidiabetic regimen of insulin and/or oral antidiabetic agents
  Other Names: Afrezza
  Arms: Technosphere® Insulin (Asthma); Technosphere® Insulin (COPD)
Drug: Usual Care — Type 1 diabetics: long-acting (basal) insulin plus rapid-acting insulin, or pre-mix insulin Type 2 diabetics: oral anti-diabetic medications with or without long-acting (basal) insulin
  Arms: Usual Care (Asthma); Usual Care (COPD)

SUMMARY:
Examine the effects of TI in combination with an anti-diabetic regimen including inhaled insulin versus anti-diabetic treatment without inhaled insulin on lung function & pulmonary safety

ELIGIBILITY:
Inclusion Criteria:

Asthma

* Physician diagnosis of asthma with history of any or all of the following: recurrent wheezing, recurrent chest tightness, recurrent difficulty breathing, or cough, particularly worse at nighttime
* Never smoked or former smokers (= 6 months since cessation)
* ≥18 years of age
* Prebronchodilator Forced Expiratory Volume in 1sec (FEV1) ≥ 60% Third National Health and Nutrition Examination Survey (NHANES III) predicted, prebronchodilator total lung capacity (TLC) ≥ 80% predicted Intermountain Thoracic Society (ITS), and prebronchodilator single breath carbon monoxide diffusing capacity of the lung (DLco) (unc) ≥70% predicted (Miller)
* < 30% day-to-day variability in daily morning Peak expiratory Volume (PEF) during the 2-week run-in period
* Significant improvement in pre- to postbronchodilator spirometry (defined as an increase from baseline of ≥ 12% and ≥ 200 mL in FEV1 or Forced Vital Capacity [FVC]) at Screening/Visit 1 or documented significant improvement in pre- to postbronchodilator spirometry (as defined above) within past 12 months in subject's medical records or a documented positive methacholine challenge test within the past 12 months

COPD

* Physician diagnosis of COPD (including emphysema and/or chronic bronchitis), history of dyspnea and/or intermittent or daily chronic cough with or without sputum production, not attributable to any other known cause
* Former smoker (≥ 6 months since cessation) with smoking history of ≥ 10 pack years
* ≥40 years of age
* Postbronchodilator FEV1/FVC ratio < 70%
* Postbronchodilator FEV1 ≥ 50% NHANES III predicted, total lung capacity (TLC) ≥ 80% predicted ITS, and DLco (unc) ≥ 50% predicted (Miller)

Both

* Clinical diagnosis of Type1 or 2 diabetes mellitus for ≥ 12 months and no change in anti-diabetic regiment for at least 90-days prior to screening
* BMI of, < 39 kg/m2
* Urine cotinine level ≤ 100ng/dL
* Clinical diagnosis of obstructive lung disease
* HbA1C > 6.5% ≤ 11.5%

Exclusion Criteria:

* History of pulmonary exacerbation within 8 weeks of screening/V1 or between V1 and V2
* Use of systemic corticosteroids or antibiotics for respiratory illness within 8 weeks of screening/V1 OR between V1 and V2
* Increase from baseline in the use of short-acting bronchodilator or short-acting anticholinergic agents, or the combination of the 2, by ≥6 puffs or ≥3 nebulizer treatments per day for ≥ 2 days
* Treatment with supplemental oxygen therapy, room air oxygen saturation, 94% or history of intubation or ICU admission for respiratory illness in the past 5 yrs.
* Greater than 2 hospitalizations or ER or urgent care visits or required >3 courses of systemic steroid in the past 12 months for respiratory illness
* Use of Symlin® (pramlintide acetate) within the preceding 90 days
* Two or more severe hypoglycemic episodes within 6 months of screening or episode of severe hypoglycemia between Screening and Baseline
* Previous exposure to any inhaled insulin product
* Currently using an insulin delivery pump
* Requires significant change (define as initiation of a new medication or change in the dose or frequency of the controller medications) in the asthma or COPD therapeutic regimen within 8 weeks of Screening/Visit 1 (Week -4) or between Visit 1 and Baseline/Visit 2
* Severe complications of diabetes mellitus, in the opinion of the PI or sub-investigator, including symptomatic autonomic neuropathy; disabling peripheral neuropathy; active proliferative retinopathy; nephropathy with renal failure, renal transplant and/or dialysis; history of foot ulcers; nontraumatic amputations due to gangrene; and/or vascular claudication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Mannkind Corporation
Locations (17):
- United States (11):
  - Mission Hills, California
  - San Diego, California
  - Palm Harbor, Florida
  - Flint, Michigan
  - Morehead City, North Carolina
  - Medford, Oregon
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Dallas, Texas
  - Federal Way, Washington
  - Tacoma, Washington
- Russia (4):
  - Yaroslavl, RUS
  - Kemerovo, RU
  - Moscow, RU
  - Saint Petersburg, RU
- Ukraine (2):
  - Kiev, UA
  - Kyiv, UA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 517 participants were screened in 5 countries . First participant was screened in March 2009.
Pre-assignment Details: 2 week screening period followed by a 2 week run-in period. After the screening period, 51 participants were randomized and 34 participants met eligibility criteria after the 2 week run-in period and were treated . Study was terminated based on data safety monitoring board recommendations.
Groups:
- Technosphere® Insulin (Asthma): Technosphere® Insulin Inhalation Powder in combination with an antidiabetic regimen in diabetic participants with Asthma
- Usual Care (Asthma): Usual and anti diabetic care in diabetic participants with Asthma.
- Technosphere® Insulin (COPD): Technosphere® Insulin Inhalation Powder in combination with an antidiabetic regimen in diabetic participants with Chronic Obstructive Pulmonary disease (COPD)
- Usual Care (COPD): Usual and anti diabetic care in diabetic participants with Chronic Obstructive Pulmonary disease (COPD)
Period: Overall Study
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care (Asthma) | Technosphere® Insulin (COPD) | Usual Care (COPD)
Started | 9 | 8 | 9 | 8
Completed | 0 | 1 | 0 | 1
Not Completed | 9 | 7 | 9 | 7
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 7 | 6 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who received at least one dose of study medication
Groups:
- Technosphere® Insulin (Asthma): Technosphere® Insulin Inhalation Powder in combination with an antidiabetic regimen in diabetic patients with Asthma
- Technosphere® Insulin (COPD): Technosphere® Insulin Inhalation Powder in combination with an antidiabetic regimen in diabetic patients with COPD
- Usual Care (COPD): Usual and anti diabetic care in diabetic participants with COPD.
- Total: Total of all reporting groups
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care (Asthma) | Technosphere® Insulin (COPD) | Usual Care (COPD) | Total
Number analyzed (Participants) | 9 | 8 | 9 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.00 (7.26) | 49.75 (15.73) | 67.44 (8.38) | 68.88 (8.20) | 64.03 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 1 | 13
  Male | 3 | 4 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-bronchodilator FEV1 From Baseline to Week 52
Description: Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) is measured at the pulmonary function laboratory.
Time Frame: 52 Weeks
Population: Only two participants completed both time points (one in the Usual Care (Asthma) Arm and one in the Usual Care (COPD) Arm); data are not provided due to privacy concerns.
Groups:
- Technosphere® Insulin (COPD): Technosphere® Insulin Inhalation Powder in combination with an antidiabetic regimen in diabetic participants with COPD
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care (Asthma) | Technosphere® Insulin (COPD) | Usual Care (COPD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Asthma Exacerbation by Treatment Arm
Description: Number of participants who experienced worsening of asthma symptoms
Time Frame: Baseline to Week 52
Population: Safety population: Participants who received at least one dose of study medication. The outcome applies only to participants with underlying Asthma
Measure: Number; unit: participants
Groups:
- Usual Care With Anti-diabetic Agents (Asthma): Usual anti diabetic care in diabetic participants with Asthma
- Usual Care With Anti-diabetic Agents (COPD): Usual anti diabetic care in diabetic participants with COPD
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care With Anti-diabetic Agents (Asthma) | Technosphere® Insulin (COPD) | Usual Care With Anti-diabetic Agents (COPD)
Number analyzed (Participants) | 9 | 8 | 0 | 0
participants
  Exacerbation of Asthma | 1 | 1 |  |
  No Exacerbation of Asthma | 8 | 7 |  |

3. Secondary Outcome: Number of Participants With COPD Exacerbation by Treatment Arm
Description: Number of participants who experienced worsening of COPD symptoms
Time Frame: Baseline to Week 52
Population: Safety population: Participants who received at least one dose of study medication. The outcome applies only to participants with underlying COPD
Measure: Number; unit: participants
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care With Anti-diabetic Agents (Asthma) | Technosphere® Insulin (COPD) | Usual Care With Anti-diabetic Agents (COPD)
Number analyzed (Participants) | 0 | 0 | 9 | 8
participants
  COPD Exacerbation |  |  | 3 | 1
  No Exacerbation |  |  | 6 | 7

4. Secondary Outcome: Change in HbA1C From Baseline to Week 52
Time Frame: Baseline, week 52
Population: as for outcome 1
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care (Asthma) | Technosphere® Insulin (COPD) | Usual Care (COPD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to 30 days after the last study visit or study related procedure was performed regardless of seriousness or relationship to investigational product
Description: Analysis was done on safety population
Arm/Group | Technosphere® Insulin (Asthma) | Usual Care With Anti-diabetic Agents (Asthma) | Technosphere® Insulin (COPD) | Usual Care With Anti-diabetic Agents (COPD)
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 8/9 | 7/8 | 4/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Technosphere® Insulin (Asthma) (N=9) | Usual Care With Anti-diabetic Agents (Asthma) (N=8) | Technosphere® Insulin (COPD) (N=9) | Usual Care With Anti-diabetic Agents (COPD) (N=8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere® Insulin (Asthma) (N=9) | Usual Care With Anti-diabetic Agents (Asthma) (N=8) | Technosphere® Insulin (COPD) (N=9) | Usual Care With Anti-diabetic Agents (COPD) (N=8)
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Monocyte count increased (Investigations) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Echymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
- Early termination of trial leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.